CLINICAL TRIAL: NCT06182995
Title: Anticipating Decline and Providing Therapy (ADAPT): Post-ICU Cognitive Screening Pilot and Feasibility Randomized Controlled Trial
Brief Title: Anticipating Decline and Providing Therapy
Acronym: ADAPT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00102934; 1K23AG073529 (NIH)
Record Dates: First submitted 2023-11-30; First posted 2023-12-27 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-07

CONDITIONS: Cognitive Impairment; Dementia; Post ICU Syndrome; Critical Illness; Cognitive Impairment, Mild
Keywords: Post ICU; Post-ICU Screening; older adults; aging
MeSH Terms: conditions — Cognitive Dysfunction; Dementia; Critical Illness

STUDY DESIGN:
Intervention Model Description: Target sample size is 120 participants, randomized 1:1 to usual care or Anticipating Decline and Providing Therapy (ADAPT) arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (Active Comparator): routine clinic visits
  Interventions: Behavioral: Usual Care post-Intensive Care Unit (ICU)
- Anticipating Decline and Providing Therapy (ADAPT) care (Experimental): The program includes a routine validated cognitive screen for high-risk older adults at 6 weeks and 6 months post-ICU discharge
  Interventions: Behavioral: Anticipating Decline and Providing Therapy (ADAPT)

INTERVENTIONS:
Behavioral: Usual Care post-Intensive Care Unit (ICU) — routine clinic visits
  Other Names: routine clinic visits
  Arms: Usual Care
Behavioral: Anticipating Decline and Providing Therapy (ADAPT) — routine validated cognitive screen for high-risk older adults at 6 weeks and 6 months post-ICU discharge
  Other Names: Post-ICU cognitive screening
  Arms: Anticipating Decline and Providing Therapy (ADAPT) care

SUMMARY:
This pilot feasibility study will be a randomized control trial of usual care following Intensive Care Unit (ICU) discharge compared to the Anticipating Decline and Providing Therapy (ADAPT) screening and support intervention. The trial aims to enroll 120 older adults (age 60 or older).

DETAILED DESCRIPTION:
Anticipating Decline and Providing Therapy (ADAPT) is a program designed to support the implementation of a routine post-ICU cognitive impairment screening and support intervention. The program includes a routine validated cognitive screen for high-risk older adults at 6 weeks and 6 months post-ICU discharge. Patients with a screening assessment that may be consistent with cognitive impairment or dementia will receive additional resources including a specialized care plan developed by the Sticht Center for Healthy Aging and Alzheimer's Prevention. The specialized care plan is adapted from a health system-based dementia care intervention and designed to support post-ICU cognitive concerns. It was adapted with input from geriatrics, intensive care, and outpatient primary care clinicians. Also conducted are semi-structured interviews with 22 older adult ICU survivors and 6 primary care physicians to elicit preferences and the intervention was further adapted based on these results.

ELIGIBILITY:
Inclusion Criteria:

* Age 60 and older at time of discharge from intensive care unit
* Minimum 72 hour Intensive Care Unit stay in an ICU at Atrium Health Wake Forest Baptist
* Delirium during ICU stay as determined by positive Confusion Assessment Method (CAM)-ICU score, review of clinical - documentation, or discussion with clinical team
* Primary care provider in the Atrium Health Wake Forest system or intention to follow with Primary Care Physician in Atrium Health system
* English speaking

Exclusion Criteria:

* Death during initial hospitalization and/or discharge to Hospice
* Life-expectancy < 6 months from pre-existing illness (defined as diagnosis of metastatic cancer, cirrhosis, advanced heart failure, prior palliative care referral)
* Acute Traumatic Brain Injury
* Continued residence in skilled nursing facility or rehab that prevents ability to complete study telephone call at time of first cognitive screen attempt
* Prior history of dementia in electronic health record
* Language or communication barrier that prohibits intervention participation
* Participant cannot identify family or caregiver contact or family/caregiver unwilling to participate
* Subject or legally authorized representative (LAR) decline consent
* Unstable telephone service for contact after hospital discharge
* Primary residence outside of North Carolina

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-03-08 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants in Cognitive Screening Intervention Arm | Week 6
  Number of participants in intervention arm who complete cognitive screening at 6 weeks

SECONDARY OUTCOMES:
Change in Percentage of participants having mild cognitive impairment (MCI), probable dementia and the combination of either MCI or probable dementia | Week 28
  percentage of participants adjudicated as having mild cognitive impairment (MCI), probable dementia and the combination of either MCI or probable dementia
Change in number of Participants between those enrolled and those who were eligible but declined | Week 52
  compare pre-specified baseline characteristics (i.e., age, sex, race, ICU length of stay) between those enrolled and those who were eligible but declined
Number of eligible participants who complete specialized care plan development visit | up to week 28
  Number of eligible participants who complete specialized care plan development visit
Change in Modified Caregiver Strain Index (MCSI) Scores | Week 28
  the modified caregiver strain index will be assessed via telephone call to identified caregiver or care partner in both groups - a 13-question tool that measures strain related to care provision - Scoring is 2 points for each 'yes', and 1 point for each 'sometimes' response. The higher the score, the higher the level of caregiver strain - range of 13-26
Change in the number of hospitalizations and Emergency Department visits | Month 12
  healthcare utilization will be the number of hospitalizations and Emergency Department (ED) visits
Change in the Number of neuropsychiatric prescriptions medications | Month 12
  number of neuropsychiatric prescriptions medications will be measured using the electronic health record
Change in number of new diagnoses of dementia or mild cognitive impairment | Month 12
  new diagnosis of dementia or mild cognitive impairment will be measured using the electronic health record
Acceptability of Intervention Measure (AIM) Scores | Week 28
  The Acceptability of Intervention Measure (AIM) - Response Scale - 4 item scales. Each item will be measured on a 5 point Likert scale: 1 = Completely disagree, 2 = Disagree, 3 = Neither agree nor disagree, 4 = Agree, 5 = Completely agree - The score is calculated mean. Higher scores reflect higher measure of acceptability
Acceptability of Intervention Appropriateness Measure (IAM) Scores | Week 28
  Intervention Appropriateness Measure (IAM) - Response Scale - 4 item scales. Each item will be measured on a 5 point Likert scale: 1 = Completely disagree, 2 = Disagree, 3 = Neither agree nor disagree, 4 = Agree, 5 = Completely agree - The score is calculated mean. Higher scores reflect higher measure of appropriateness
Acceptability of Feasibility of Intervention measure (FIM) Scores | Week 28
  The Acceptability of Feasibility of Intervention Measure (FIM) - Response Scale - 4 item scales. Each item will be measured on a 5 point Likert scale: 1 = Completely disagree, 2 = Disagree, 3 = Neither agree nor disagree, 4 = Agree, 5 = Completely agree - The score is calculated mean. Higher scores reflect higher measure of feasibility

OTHER OUTCOMES:
Qualitative Perception | Week 28
  semi-structured interviews with participants for feedback about the intervention - this will not be a numerical score

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Palakshappa, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Atrium Health Wake Forest Baptist, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No